CLINICAL TRIAL: NCT00307983
Title: Effect of Malnutrition on the Prognosis in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Shizuoka (Other)
Other Study IDs: CT2006002
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-03-28 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Renal Failure; Hemodialysis; Malnutrition
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examined the effect of malnutrition and/or inflammation on atherosclerosis and prognosis in hemodialysis.

DETAILED DESCRIPTION:
Malnutrition is known to affect their prognosis in hemodialysis patients. Furthermore, recent studies indicate that malnutrition is associated with inflammation and atherosclerosis in these patients. In this study we examine the effect of malnutrition and/or inflammation on atherosclerosis and 5-year survival rate in 600 hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for at least 6 months

Exclusion Criteria:

* disabled patients

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2004-04; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Hiromichi Kumagai, MD, Study Chair — University of Shizuoka
Locations (2):
- Japan (2):
  - Maruyama Hospital, Hamamatsu, Shizuoka
  - Iwata City Hospital, Iwata, Shizuoka